CLINICAL TRIAL: NCT04824001
Title: Using Exercise Echocardiography to Investigate the Effects of Different Exercise Trainings on Left Ventricular Mechanics in Patients With Coronary Artery Disease: a Speckle-tracking Echocardiography
Brief Title: Exercise Echocardiography on LV Mechanics in Patients With CAD: a Speckle-tracking Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Other Study IDs: CMUH108-REC2-180
Record Dates: First submitted 2021-02-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases; STEMI; NSTEMI
Keywords: stress echocardiography; speckle tracking
MeSH Terms: conditions — Cardiovascular Diseases; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI: ST-segment elevation myocardial infarction (STEMI) is defined by symptoms of myocardial ischemia accompanied by a persistent elevation of the ST segment on the electrocardiogram (ECG) and the subsequent release of biomarkers of myocardial necrosis.
  Interventions: Other: exercise stress echocardiography
- NSTEMI: If there is elevation of the blood markers suggesting heart damage, but no ST elevation seen on the EKG tracing, this is known as a non ST-elevation myocardial infarction (NSTEMI).
  Interventions: Other: exercise stress echocardiography

INTERVENTIONS:
Other: exercise stress echocardiography — Stress echocardiography test. The standardized exercise test was conducted by 50-W semi-recumbent cycling for 3 min. Stress echocardiograph images were acquired at the third minute of cycling to ensure that subjects had reached a steady-state HR.

SUMMARY:
Recovering blood flow to a coronary stenosis may improve left ventricular (LV) function in patients with coronary artery disease (CAD). However, the reported data about evaluation of LV function post-percutaneous coronary intervention (PCI) in CAD was limited. The aim of this study was to compare the LV function measured by 3 min low dose exercise stress echocardiography (ESE) combined 2D speckle tracking echocardiography (STE) in patients with CAD underwent PCI, and to identify factors affecting the change of LV function. Patients with CAD who underwent acute PCI were enrolled.

DETAILED DESCRIPTION:
The assessment of temporal changes in systolic and diastolic regional left ventricle function by 2D-STE after successful reperfusion therapy of acute myocardial infarction (AMI).The estimated total number of participants is 90 patients with AMI and treated with successful percutaneous coronary intervention were included in this study. The echocardiographic measurements were performed in all patients within in-hotpital after PCI procedure, and then followed up at 7, 14, 30, 60 and 180 days after discharge. Recovery of regional systolic and diastolic myocardial function after acute myocardial infarction evaluated by ESE-STE.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction diagnosed by a physician
* undergoing percutaneous coronary intervention
* Exercise testing and stress echocardiography are performed with the approval of the physician.

Exclusion Criteria:

* Severe cardiac valve disease
* Left bundle branch block
* Uncontrolled diabetes or hypertension
* Orthopedics or other conditions that hinder from exercise
* Uncontrolled sinus tachycardia (greater than 120 beats per minute)

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: acute myocardial infarction diagnosed by a physician and undergoing percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
The alterations of LV mechanics responses to a 3-min low dose exercise stress echocardiography following time. | detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.
  The STE was performed at rest, during exercise and recovery to compare the changes of LV machines following discharge. The standardized exercise test was conducted by 50-W semirecumbent cycling (Cardiac Stress Table w/Angio) for 3 min. Stress echocardiograph images were acquired at the third minute of cycling to ensure that subjects had reached a steady-state HR.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | detected at the day 30, 60, and 180 after discharge.
  The graded exercise test (GXT) was performed with a cycle ergometer at the day 30 and 180 after discharge. The GXT comprised of unloaded pedaling for 2 min followed by a continuous increase in work rate (20-30 W) every 3 min until exhaustion (i.e., V˙ O2max). Minute ventilation (V˙ E), V˙ O2, and CO2 production (V˙ CO2) were measured breath-by-breath using a computer-based system (MasterScreen CPX; Cardinal Health Germany).
The brain-type natriuretic peptide (BNP) levels | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  BNP levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
The high-sensitivity CRP (hsCRP) levels | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  hsCRP levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
The creatine kinase (CK) levels | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  The CK levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
The creatine kinase-MB (CK-MB) levels | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  The CK-MB levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
The troponin I levels | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  The troponin I levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
The left ventricle wall and cavity dimensions | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  M-mode images were used to determine the LV wall and cavity dimensions at end-systole and end-diastole from a parasternal long axis view.
The left ventricle mass | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  Measurements of LVmass and the short fraction index were automatically derived using standard equations as followed: LVmass(gm) = 0.77 X 10^-3X [(IVS + LVIDd +PW)^3 - (LVIDd)^3 + 2.4]
The left ventricle ejection fraction | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  LV ejection fraction (LVEF) was determined using the modified Simpson's method from the apical four-chamber views.
The left ventricle diastolic functions | detected at the detected at the in-hospital and the day 7, 14, 30, 60, and 180 after discharge.ay 30, 60, and 180 after discharge.
  Analysis of Doppler pulsed wave was performed to determine diastolic transmitral blood flow velocities for peak early (E) and late (A) fillings and was also detected the diastolic mitral annular tissue velocities for peak early (E') and late (A') fillings.

CONTACTS AND LOCATIONS:
Overall Officials: LI-Wei Chou, PhD, Principal Investigator — China Medical University Hospital/Asia University Hospital
Locations (1):
- Asia University Hospital, Wufeng District, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anand IS, Kuskowski MA, Rector TS, Florea VG, Glazer RD, Hester A, Chiang YT, Aknay N, Maggioni AP, Opasich C, Latini R, Cohn JN. Anemia and change in hemoglobin over time related to mortality and morbidity in patients with chronic heart failure: results from Val-HeFT. Circulation. 2005 Aug 23;112(8):1121-7. doi: 10.1161/CIRCULATIONAHA.104.512988. Epub 2005 Aug 15. PMID 16103233
- [Background] Sikora-Frac M, Zaborska B, Maciejewski P, Budaj A, Bednarz B. Improvement of left ventricular function after percutaneous coronary intervention in patients with stable coronary artery disease and preserved ejection fraction: Impact of diabetes mellitus. Cardiol J. 2021;28(6):923-931. doi: 10.5603/CJ.a2019.0066. Epub 2019 Jul 1. PMID 31257568
- [Background] Li H, Liu C, Zhang G, Wang C, Sun P, Du G, Tian J. The early alteration of left ventricular strain and dys-synchrony index in breast cancer patients undergoing anthracycline therapy using layer-specific strain analysis. Echocardiography. 2019 Sep;36(9):1675-1681. doi: 10.1111/echo.14460. Epub 2019 Aug 27. PMID 31454106
- [Background] Huang YC, Tsai HH, Fu TC, Hsu CC, Wang JS. High-Intensity Interval Training Improves Left Ventricular Contractile Function. Med Sci Sports Exerc. 2019 Jul;51(7):1420-1428. doi: 10.1249/MSS.0000000000001931. PMID 30829901